CLINICAL TRIAL: NCT05793463
Title: Anti-mullerian Hormone in Pediatric Patients Treated for Acute Lymphoblastic Leukemia
Brief Title: Anti-mullerian Hormone in Acute Lymphoblastic Leukemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 03/17
Record Dates: First submitted 2023-03-20; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia; Fertility preservation; Anti-Mullerian hormone
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute lymphoblastic leukemia (ALL) is the most common childhood malignancy, with current survival rates exceeding 90%. As cure rates improve, increasing attention is focused on survivor quality of life, including fertility. It is generally accepted that cancer treatments in childhood may interfere with gonadal function, reducing the pool of primordial follicles and consequently causing premature menopause in women. Anti-Mullerian hormone (AMH) levels is a valuable quantitative indicator of ovarian reserve, being directly related to the number of antral follicles. The evaluation of this hormone makes it possible to identify women at risk of early menopause and to propose them interventions for monitoring and preservation of oocytes, allowing girls to be able to have children once they reach adulthood. The objective of this study is to determine ovarian reserve in girls with ALL before and after treatment by means of the evaluation of the AMH assay.

ELIGIBILITY:
Inclusion Criteria:

* Female less than 18 years of age
* Diagnosis of acute lymphoblastic leukemia
* enrollment within the first month after diagnosis

Exclusion Criteria:

* Previous treatments with cytostatics drugs
* ALL as a second malignancy
* Syndromic patient or primary hypogonadism

Ages: 1 Month to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Female less than 18 years of age with ALL
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2018-02-15 (Actual); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Evaluation of blood AMH levels before ALL treatment | Within one months from ALL diagnosis
  AMH levels will be evaluated in peripheral blood
Evaluation of blood AMH levels after ALL treatment | 24 months after ALL diagnosis
  AMH levels will be evaluated in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Nagua Giurici, MD, Study Director — IRCCS materno infantile Burlo Garofolo
Locations (1):
- IRCCS Burlo Garofolo, Trieste, Italy